CLINICAL TRIAL: NCT04676399
Title: Improving Pain Management Via Spinal Cord Stimulation and Blood Pressure Reduction (PASSION Study)
Brief Title: Improving Pain Management Via Spinal Cord Stimulation and Blood Pressure Reduction
Acronym: PASSION
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 00146604
Record Dates: First submitted 2020-11-19; First posted 2020-12-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Hypertension; Diuretics Drug Reactions; SCS
MeSH Terms: conditions — Chronic Pain; Hypertension | interventions — Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: Mixed Model 2-way analysis of variance to asses pain and BP responses to the diuretic vs. placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization to either hydrochlorothiazide or placebo using a crossover study design will occur via a 1:1 ratio determined by computer generated randomization
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydrochlorothiazide Pill (12.5 mg twice a day) (Experimental): Planned use in this study
  1. Condition/disease indication(s): Hypertension
  2. Subject population: Chronic pain
  3. Dose(s): 12.5 mg twice per day for 14 days.
  4. Administration: Oral
  5. Dosing regimen: 12.5 mg twice per day
  Interventions: Drug: Hydrochlorothiazide 12.5mg
- Placebo (Placebo Comparator): Has no active ingredients but is made to look like the study drug.
  2 pills/day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrochlorothiazide 12.5mg — 2 pills/day (1 pill every morning and 1 pill every evening) for 14 days.
  Other Names: HCTZ
  Arms: Hydrochlorothiazide Pill (12.5 mg twice a day)
Drug: Placebo — 2 pills/day (1 pill every morning and 1 pill every evening) for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study (PASSION study) is to monitor symptoms of chronic pain before and after 2 weeks of a standard drug commonly used to treat elevated blood pressure compared with 2 weeks of placebo (crossover design) so that we may better understand how blood pressure affects your level of pain. This study is not testing an experimental drug.

DETAILED DESCRIPTION:
The goal of the PASSION study is to determine the extent to which reductions in blood pressure improve pain management via SCS

1. Examine the extent to which reductions in blood pressure (2 weeks of diuretic and 2 weeks of placebo) improve pain management among patients with chronic pain and hypertension compared.
2. Examine the extent to which arterial baroreflex function, which is critical to blood pressure regulation, is impaired in patients with chronic pain and hypertension and is correlated with chronic pain symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, age 40-79
2. Chronic low back pain
3. Permanent spinal cord stimulator implant for chronic pain
4. Stage 1 hypertension (BP 130-139/80-89 mmHg) with ASCVD risk ≥10%
5. Stage 2 hypertension (BP ≥ 140/90 mmHg)
6. Willing to visit research lab (Fairway CTSU)
7. Willing to undergo a blood draw
8. Able to provide written informed consent

Exclusion Criteria:

1. Any history of abnormal responses (allergy) to thiazide-type drugs
2. Currently taking any antihypertensive medication
3. Stage 1 hypertension (BP 130-139/80-89 mmHg) with ASCVD risk <10%
4. BP ≥160/100 (these patients should be promptly treated with 2 medications)
5. Secondary hypertension (e.g., aldosteronism, renal artery stenosis)
6. Symptomatic hypotension (weakness or syncope upon standing)
7. Renal failure
8. Diabetes requiring insulin or glucose-lowering drugs
9. History of neurological disease (e.g., dementias, Parkinson's)
10. History of stroke
11. Current diagnosis of cancer
12. Women who are pregnant or planning to become pregnant
13. Any active infection
14. Subject is unwilling or unable to comply with the protocol
15. If currently taking a NSAID, willing to stop for at least 3 days prior to beginning study and throughout study

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure Measurement From Visit 1 to Visit 2 | 1 week
  Measurements of blood pressure via arm cuff and finger cuff
Change in Blood Pressure Measurement From Visit 2 to Visit 3 | 1 week
  Measurements of blood pressure via arm cuff and finger cuff
Change in Blood Pressure Measurement From Visit 3 to Visit 4 | 1 week
  Measurements of blood pressure via arm cuff and finger cuff
Change in Blood Pressure Measurement From Visit 4 to Visit 5 | 2 week
  Measurements of blood pressure via arm cuff and finger cuff
Change from Visit 1 PainDETECT Questionnaire to Visit 2 | 1 week
  A battery of questionnaires is intended to understand key aspects of pain, mood, and function as quickly and efficiently as possible. The focus of these measures is on obtaining an accurate assessment of pain, while also asking about physical function, anxiety, and other associated somatic disturbances. These questionnaires will be taken prior to SCS implant (Baseline) and after SCS implant (1 week post-op, 4 weeks post-op, and 8 weeks post-op ) to assess and compare.
  Neuropathic Pain Descriptors: The Pain DETECT is a 9-item measure of sensory descriptors and spatial and temporal characteristics that has demonstrated utility in identifying central neuropathic pain.
Change from Visit 2 PainDETECT Questionnaire to Visit 3 | 1 week
  A battery of questionnaires is intended to understand key aspects of pain, mood, and function as quickly and efficiently as possible. The focus of these measures is on obtaining an accurate assessment of pain, while also asking about physical function, anxiety, and other associated somatic disturbances. These questionnaires will be taken prior to SCS implant (Baseline) and after SCS implant (1 week post-op, 4 weeks post-op, and 8 weeks post-op ) to assess and compare.
  Neuropathic Pain Descriptors: The Pain DETECT is a 9-item measure of sensory descriptors and spatial and temporal characteristics that has demonstrated utility in identifying central neuropathic pain.
Change from Visit 3 PainDETECT Questionnaire to Visit 4 | 1 week
  A battery of questionnaires is intended to understand key aspects of pain, mood, and function as quickly and efficiently as possible. The focus of these measures is on obtaining an accurate assessment of pain, while also asking about physical function, anxiety, and other associated somatic disturbances. These questionnaires will be taken prior to SCS implant (Baseline) and after SCS implant (1 week post-op, 4 weeks post-op, and 8 weeks post-op ) to assess and compare.
  Neuropathic Pain Descriptors: The Pain DETECT is a 9-item measure of sensory descriptors and spatial and temporal characteristics that has demonstrated utility in identifying central neuropathic pain.
Change from Visit 4 PainDETECT Questionnaire to Visit 5 | 2 week
  A battery of questionnaires is intended to understand key aspects of pain, mood, and function as quickly and efficiently as possible. The focus of these measures is on obtaining an accurate assessment of pain, while also asking about physical function, anxiety, and other associated somatic disturbances. These questionnaires will be taken prior to SCS implant (Baseline) and after SCS implant (1 week post-op, 4 weeks post-op, and 8 weeks post-op ) to assess and compare.
  Neuropathic Pain Descriptors: The Pain DETECT is a 9-item measure of sensory descriptors and spatial and temporal characteristics that has demonstrated utility in identifying central neuropathic pain.
Visit 1 Catecholamines( Norepinephrine) & Tumor necrosis factor-alpha (TNF-α) and interlukin-6 (IL6) Blood Work | Visit 1 (Day 1)
  Catecholamines( Norepinephrine) Blood Test: pg/mL
  • normal range for norepinephrine is 70 to 1700 pg/mL
  Tumor necrosis factor-alpha (TNF-α) and interlukin-6 (IL6) Blood Test: pg/mL
  * IL-6 normal values was 6-31 pg/mL
  * TNF-α 5 pg/mL,
Visit 1 Lipid Panel Blood Work Results | Visit 1 (Day 1)
  Lipid panel Blood Test: mg/dL,
  * Total Cholesterol Less than 170mg/dL
  * Non-HDL Less than 120mg/dL
  * LDL Less than 100mg/dL
  * HDL More than 45mg/dL
Visit 1 Comprehensive Metabolic Panel Blood Work Results | Visit 1 (Day 1)
  Metabolic Panel Blood Test (Electrolyte Check): mg/dL, mmol/L , g/dL, U/L, mEq/L
  * Albumin: 3.4 to 5.4 g/dL (34 to 54 g/L)
  * Alkaline phosphatase: 20 to 130 U/L
  * ALT (alanine aminotransferase): 4 to 36 U/L
  * AST (aspartate aminotransferase): 8 to 33 U/L
  * BUN (blood urea nitrogen): 6 to 20 mg/dL (2.14 to 7.14 mmol/L)
  * Calcium: 8.5 to 10.2 mg/dL (2.13 to 2.55 mmol/L)
  * Chloride: 96 to 106 mEq/L (96 to 106 mmol/L)
  * CO2 (carbon dioxide): 23 to 29 mEq/L (23 to 29 mmol/L)
  * Creatinine: 0.6 to 1.3 mg/dL (53 to 114.9 µmol/L)
  * Glucose: 70 to 100 mg/dL (3.9 to 5.6 mmol/L)
  * Potassium: 3.7 to 5.2 mEq/L (3.70 to 5.20 mmol/L)
  * Sodium: 135 to 145 mEq/L (135 to 145 mmol/L)
  * Total bilirubin: 0.1 to 1.2 mg/dL (2 to 21 µmol/L)
  * Total protein: 6.0 to 8.3 g/dL (60 to 83 g/L)
Visit 1 Stored Plasma Blood Work Results | Visit 1 (Day 1)
  Stored plasma for inflammatory markers
Visit 2 Comprehensive Metabolic Panel/Electrolyte Check Blood Work Results | Visit 2 (Day 7)
  Metabolic Panel Blood Test (Electrolyte Check): mg/dL, mmol/L , g/dL, U/L, mEq/L
  * Albumin: 3.4 to 5.4 g/dL (34 to 54 g/L)
  * Alkaline phosphatase: 20 to 130 U/L
  * ALT (alanine aminotransferase): 4 to 36 U/L
  * AST (aspartate aminotransferase): 8 to 33 U/L
  * BUN (blood urea nitrogen): 6 to 20 mg/dL (2.14 to 7.14 mmol/L)
  * Calcium: 8.5 to 10.2 mg/dL (2.13 to 2.55 mmol/L)
  * Chloride: 96 to 106 mEq/L (96 to 106 mmol/L)
  * CO2 (carbon dioxide): 23 to 29 mEq/L (23 to 29 mmol/L)
  * Creatinine: 0.6 to 1.3 mg/dL (53 to 114.9 µmol/L)
  * Glucose: 70 to 100 mg/dL (3.9 to 5.6 mmol/L)
  * Potassium: 3.7 to 5.2 mEq/L (3.70 to 5.20 mmol/L)
  * Sodium: 135 to 145 mEq/L (135 to 145 mmol/L)
  * Total bilirubin: 0.1 to 1.2 mg/dL (2 to 21 µmol/L)
  * Total protein: 6.0 to 8.3 g/dL (60 to 83 g/L)
Visit 3 Comprehensive Metabolic Panel/Electrolyte Check Blood Work Results | Visit 3 (Day 14)
  Metabolic Panel Blood Test (Electrolyte Check): mg/dL, mmol/L , g/dL, U/L, mEq/L
  * Albumin: 3.4 to 5.4 g/dL (34 to 54 g/L)
  * Alkaline phosphatase: 20 to 130 U/L
  * ALT (alanine aminotransferase): 4 to 36 U/L
  * AST (aspartate aminotransferase): 8 to 33 U/L
  * BUN (blood urea nitrogen): 6 to 20 mg/dL (2.14 to 7.14 mmol/L)
  * Calcium: 8.5 to 10.2 mg/dL (2.13 to 2.55 mmol/L)
  * Chloride: 96 to 106 mEq/L (96 to 106 mmol/L)
  * CO2 (carbon dioxide): 23 to 29 mEq/L (23 to 29 mmol/L)
  * Creatinine: 0.6 to 1.3 mg/dL (53 to 114.9 µmol/L)
  * Glucose: 70 to 100 mg/dL (3.9 to 5.6 mmol/L)
  * Potassium: 3.7 to 5.2 mEq/L (3.70 to 5.20 mmol/L)
  * Sodium: 135 to 145 mEq/L (135 to 145 mmol/L)
  * Total bilirubin: 0.1 to 1.2 mg/dL (2 to 21 µmol/L)
  * Total protein: 6.0 to 8.3 g/dL (60 to 83 g/L)
Visit 4 Comprehensive Metabolic Panel/Electrolyte Check Blood Work Results | Visit 4 (Day 21)
  Metabolic Panel Blood Test (Electrolyte Check): mg/dL, mmol/L , g/dL, U/L, mEq/L
  * Albumin: 3.4 to 5.4 g/dL (34 to 54 g/L)
  * Alkaline phosphatase: 20 to 130 U/L
  * ALT (alanine aminotransferase): 4 to 36 U/L
  * AST (aspartate aminotransferase): 8 to 33 U/L
  * BUN (blood urea nitrogen): 6 to 20 mg/dL (2.14 to 7.14 mmol/L)
  * Calcium: 8.5 to 10.2 mg/dL (2.13 to 2.55 mmol/L)
  * Chloride: 96 to 106 mEq/L (96 to 106 mmol/L)
  * CO2 (carbon dioxide): 23 to 29 mEq/L (23 to 29 mmol/L)
  * Creatinine: 0.6 to 1.3 mg/dL (53 to 114.9 µmol/L)
  * Glucose: 70 to 100 mg/dL (3.9 to 5.6 mmol/L)
  * Potassium: 3.7 to 5.2 mEq/L (3.70 to 5.20 mmol/L)
  * Sodium: 135 to 145 mEq/L (135 to 145 mmol/L)
  * Total bilirubin: 0.1 to 1.2 mg/dL (2 to 21 µmol/L)
  * Total protein: 6.0 to 8.3 g/dL (60 to 83 g/L)
Visit 5 Comprehensive Metabolic Panel/Electrolyte Check Blood Work Results | Visit 5 (Day 28)
  Metabolic Panel Blood Test (Electrolyte Check): mg/dL, mmol/L , g/dL, U/L, mEq/L
  * Albumin: 3.4 to 5.4 g/dL (34 to 54 g/L)
  * Alkaline phosphatase: 20 to 130 U/L
  * ALT (alanine aminotransferase): 4 to 36 U/L
  * AST (aspartate aminotransferase): 8 to 33 U/L
  * BUN (blood urea nitrogen): 6 to 20 mg/dL (2.14 to 7.14 mmol/L)
  * Calcium: 8.5 to 10.2 mg/dL (2.13 to 2.55 mmol/L)
  * Chloride: 96 to 106 mEq/L (96 to 106 mmol/L)
  * CO2 (carbon dioxide): 23 to 29 mEq/L (23 to 29 mmol/L)
  * Creatinine: 0.6 to 1.3 mg/dL (53 to 114.9 µmol/L)
  * Glucose: 70 to 100 mg/dL (3.9 to 5.6 mmol/L)
  * Potassium: 3.7 to 5.2 mEq/L (3.70 to 5.20 mmol/L)
  * Sodium: 135 to 145 mEq/L (135 to 145 mmol/L)
  * Total bilirubin: 0.1 to 1.2 mg/dL (2 to 21 µmol/L)
  * Total protein: 6.0 to 8.3 g/dL (60 to 83 g/L)
Visit 5 Lipid Panel Blood Work Results | Visit 5 (Day 28)
  Lipid panel Blood Test: mg/dL,
  * Total Cholesterol Less than 170mg/dL
  * Non-HDL Less than 120mg/dL
  * LDL Less than 100mg/dL
  * HDL More than 45mg/dL
Visit 5 Stored Plasma Blood Work Results | Visit 5 (Day 35)
  Stored plasma for inflammatory markers Blood Test
Visit 5 Catecholamines( Norepinephrine) & Tumor necrosis factor-alpha (TNF-α) and interlukin-6 (IL6) Blood Work | Visit 5 (Day 28)
  Catecholamines( Norepinephrine) Blood Test: pg/mL
  • normal range for norepinephrine is 70 to 1700 pg/mL
  Tumor necrosis factor-alpha (TNF-α) and interlukin-6 (IL6) Blood Test: pg/mL
  * IL-6 normal values was 6-31 pg/mL
  * TNF-α 5 pg/mL,

CONTACTS AND LOCATIONS:
Overall Officials: Seth W Holwerda, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The Marc A. Asher Comprehensive Spine Center at the Kansas University Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be available upon reasonable request